CLINICAL TRIAL: NCT06615752
Title: A Phase I/II Study to Determine the Safety and Efficacy of a Combination of Green Tea and Quercetin With Docetaxel in Castration-resistant Prostate Cancer Patients
Brief Title: Green Tea and Quercetin in Combination With Docetaxel Chemotherapy in Castration-resistant Prostate Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Watts Healthcare Corporation (Unknown)
Responsible Party: Principal Investigator, Piwen Wang, Associate Professor, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2188250-3; 2U54MD007598-16 (NIH)
Record Dates: First submitted 2024-09-16; First posted 2024-09-27 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC)
Keywords: green tea; quercetin; docetaxel; prostate cancer; phase II
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tea; Quercetin; Docetaxel

STUDY DESIGN:
Intervention Model Description: This study includes a dose-escalation study and an expanded phase II study. For the dose-escalation study, patients will be assigned to different dose levels in the order of recruiting. For the expanded phase II study, patients will be randomly assigned to the green tea plus quercetin group receiving green tea + quercetin + docetaxel, or the placebo group receiving placebo + docetaxel.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- green tea and quercetin (Experimental): Green tea and quercetin capsules will be administered in combination with docetaxel treatment.
  Interventions: Drug: green tea and quercetin + docetaxel
- placebo (Placebo Comparator): Placebo capsules will be administered in combination with docetaxel treatment as comparison.
  Interventions: Drug: Placebo + docetaxel

INTERVENTIONS:
Drug: green tea and quercetin + docetaxel — green tea and quercetin supplements in combination with docetaxel infusion
  Other Names: GT and Q
  Arms: green tea and quercetin
Drug: Placebo + docetaxel — Placebo will be given along with docetaxel chemotherapy
  Other Names: Placebo
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to find out if taking natural products green tea and quercetin along with docetaxel chemotherapy improves the therapy of advanced prostate cancer, i.e., metastatic castration-resistant prostate cancer (mCRPC). It will also learn about the safety of this combination.

Researchers will compare green tea plus quercetin to a placebo (a look-alike substance that contains no drug) in combination with docetaxel to see if green tea and quercetin works to improve the therapeutic effect of docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form and HIPPA (Health Insurance Portability and Accountability Act) authorization.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male patients 18 years or older
* Diagnosed with metastatic prostate cancer
* History of confirmed progressive disease with concurrent use of medical castration (e.g. luteinizing hormone-releasing hormone analogue), or surgical castration
* Confirmed progressive disease with concurrent use of enzalutamide, apalutamide, darolutamide, and/or abiraterone acetate
* Clinical decision to start doc infusion with prednisone treatment
* Adequate bone marrow function (absolute neutrophil count (ANC) more than1500 cells/mm³, platelet count more than 100,000 cells/mm³)
* Adequate liver function (total bilirubin less than upper limit of normal (ULN), alanine aminotransferase (ALT) less than 1.5 x ULN, aspartate aminotransferase (AST) less than 1.5 x ULN)
* Adequate renal function (serum creatinine level within normal limits)
* At least a 6-month or greater life expectancy
* Willing to stop consuming tea or tea-containing products and quercetin supplements throughout the entire intervention period except for the green tea extract and quercetin provided during study intervention

Exclusion Criteria:

* Prior treatment of chemotherapy and/or radiotherapy for metastatic disease
* Any comorbid condition that would preclude the administration of docetaxel/prednisone
* Ongoing alcohol abuse
* Significant medical or psychiatric conditions that would make the patient a poor protocol candidate
* Prior allergic reaction to tea, tea products or quercetin supplements
* Allergies to multiple food items or nutritional supplements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only biologically male is eligible for this study
Enrollment: 99 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy evaluated with blood prostate specific antigen (PSA) level | From enrollment to the end of treatment at 11 weeks
  Blood PSA will be measured at baseline, 1st day of each cycle of docetaxel treatment (21 days per cycle, for 3 cycles), and at the end of the intervention.

SECONDARY OUTCOMES:
circulating tumor DNA level (ctDNA) analyzed by next generation sequencing | From the start of intervention at 3 weeks to the end of treatment at 11 weeks.
  CtDNA will be measured at the 1st day of each cycle of docetaxel treatment, and at the end of the intervention.
tumor burden by CT detection | From the start of intervention at 3 weeks to the end of treatment at 11 weeks.
  Tumor burden, including tumor number and size, will be assessed in both primary and metastatic sites using computed tomography (CT), to assist in the evaluation of complete response vs. stable disease vs. progressive disease using the RECIST criteria.
Adverse events graded by using NCI CTCAE criteria | From the start of intervention at 3 weeks to the end of treatment at 11 weeks.
  The Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, will be followed for a comprehensive evaluation of adverse events in multiple systems including blood, liver, gastrointestinal tract, and neural system.
Area under curve (AUC) of blood green tea, quercetin, and docetaxel | On the 1st day of cycle 1 (each cycle is 21 days, 3 cycles total) of the dose escalation study.
  The AUC of blood green tea, quercetin, and docetaxel will be analyzed in cycle 1 of different dose levels in the dose escalation study.
Maximum concentrations (Cmax) of blood green tea, quercetin, and docetaxel | On the 1st day of cycle 1 (each cycle is 21 days, 3 cycles total) of the dose escalation study.
  The Cmax of blood green tea, quercetin, and docetaxel will be analyzed in cycle 1 of different dose levels in the dose escalation study.
Time taken to reach the maximum concentration (Tmax) | On the 1st day of cycle 1 (each cycle is 21 days, 3 cycles total) of the dose escalation study.
  The Tmax of blood green tea, quercetin, and docetaxel will be analyzed in cycle 1 of different dose levels in the dose escalation study.

CONTACTS AND LOCATIONS:
Overall Officials: Piwen Wang, PhD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles R. Drew University of Medicine and Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No